CLINICAL TRIAL: NCT06686459
Title: A Single-center Prospective Phase II Clinical Study With a Non-blind, Single-arm Design Combined With a Parallel External Control Group to Evaluate the Efficacy and Safety of Artificial Intelligence-assisted One-stop Radiotherapy After Breast-conserving Surgery
Brief Title: A Phase II Clinical Trial of Artificial Intelligence-assisted One-stop Radiotherapy for Breast Cancer After Breast-conserving Surgery
Acronym: BC-AIO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Wei-Hong Zheng, Principal Investigator, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SL-B2024-438-03
Record Dates: First submitted 2024-11-06; First posted 2024-11-13 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer Invasive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ALL-in-one group (Experimental): ALL-in-one radiotherapy (breast + supraclavicular + internal mammary lymph node drainage area)
  Interventions: Radiation: ALL-in-one radiotherapy
- IMRT group (Placebo Comparator): IMRT (breast + supraclavicular + internal mammary lymph node drainage area)
  Interventions: Radiation: IMRT

INTERVENTIONS:
Radiation: ALL-in-one radiotherapy — ALL-in-one radiotherapy (breast + supraclavicular + internal mammary lymph node drainage area)
  Arms: ALL-in-one group
Radiation: IMRT — IMRT (breast + supraclavicular + internal mammary lymph node drainage area)
  Arms: IMRT group

SUMMARY:
Background: Breast cancer became the most prevalent cancer globally in 2020, and post-surgery radiotherapy is crucial for most patients. Traditional radiotherapy is complex and time-consuming, affecting patient experience. To streamline this, an AI-assisted All-in-one (AIO) radiotherapy approach has been developed, integrating steps like target delineation and planning to reduce wait times and enhance accuracy. Preliminary results are promising, with significant time savings and high pass rates in initial assessments. Further exploration is needed to confirm the accuracy, effectiveness, and safety of AIO radiotherapy.

Primary objective: To conduct a prospective phase II clinical trial to determine the feasibility (including efficacy and safety) of AIO radiotherapy, and to provide a basis for establishing standard operating procedures.

Secondary objectives: To assess the impact of AIO radiotherapy on overall survival, local regional recurrence, and distant metastasis rates. To investigate the incidence and contributing factors of cardiac damage after AIO radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* 1. Female patients aged 18-70 years. 2. ECOG performance status of 0-2. 3. Newly diagnosed invasive breast cancer, underwent breast-conserving surgery plus axillary lymph node dissection, with positive axillary lymph nodes (ypN+) and negative surgical margins.

  4. No distant metastasis. 5. Capable of tolerating radiotherapy. 6. For ER/PR-positive patients, willing to receive anticipated 5 years of endocrine therapy.

  7. For HER2-positive patients, willing to receive anticipated 1 year of anti-HER2 targeted therapy.

  8. For patients requiring neoadjuvant/adjuvant chemotherapy, must have completed chemotherapy.

  9. Left ventricular ejection fraction (LVEF) measured by echocardiography is 50%.

  10. Must undergo adjuvant IMRT (Intensity-Modulated Radiation Therapy). 11. Capable of tolerating lying still on the treatment accelerator bed for 30 minutes to complete All-In-One radiotherapy.

  12. Have follow-up conditions and are willing to adhere to follow-up. 13. Signed an informed consent form.

Exclusion Criteria:

* 1. Synchronous bilateral breast cancer; sentinel lymph node biopsy of the axilla was performed without axillary lymph node dissection.

  2. Stage I breast reconstruction surgery or expander implantation surgery on the affected side chest wall.

  3. The purpose of radiotherapy is palliative. 4. Myocardial infarction within the last 3 months or uncorrected unstable arrhythmia or uncorrected unstable angina.

  5. History of chest wall or supraclavicular radiotherapy in the past; past or concurrent second primary malignant tumors (except for non-melanoma skin cancer, papillary/follicular thyroid carcinoma, and carcinoma in situ of the cervix).

  6. All-in-one one-stop radiotherapy has not been completed.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 860 (Estimated)
Dates: Start 2025-04-06 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
incidence rate of adverse effects | 12 months after the end of radiotherapy

SECONDARY OUTCOMES:
overall survical | measured from baseline through study completion, an average of 1 year
disease free survival | measured from baseline through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No